CLINICAL TRIAL: NCT02274818
Title: Individualized Comparative Effectiveness of Models Optimizing Patient Safety and Resident Education (iCOMPARE).
Brief Title: Individualized Comparative Effectiveness of Models Optimizing Patient Safety and Resident Education.
Acronym: iCOMPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Johns Hopkins University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00051227; 1U01HL125388 (NIH); 1U01HL126088 (NIH)
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Safety; Education, Medical; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Duty Hour Schedule (No Intervention): IM programs randomized to the currently mandated duty 16 hour standards (maximum work duration of 16 hours for interns and 28 hours for PGY2-3); this schedule may involve night float.
- Flexible Duty Hour Schedule (Experimental): IM programs randomized to intervention will be allowed to construct flexible duty hour schedules that comply with 3 rules:
  * No more than 80 hours of work per week (when averaged over 4 weeks)
  * 1 day off in 7 (when averaged over 4 weeks)
  * In-house call no more frequently than every 3rd night (when averaged over 4 weeks)
  Interventions: Behavioral: Flexible Duty Hour Schedule

INTERVENTIONS:
Behavioral: Flexible Duty Hour Schedule — IM programs randomized to intervention will be allowed to construct flexible duty hour schedules that comply with 3 rules:
  * No more than 80 hours of work per week (when averaged over 4 weeks)
  * 1 day off in 7 (when averaged over 4 weeks)
  * In-house call no more frequently than every 3rd night (when averaged over 4 weeks)
  Arms: Flexible Duty Hour Schedule

SUMMARY:
The investigators are conducting a cluster randomized trial in a sample of 63 internal medicine (IM) training programs that are randomly assigned to either the current duty hour standards or less restricted flexible duty hour standards.

The trial includes a main protocol in which all randomized IM programs participate and two substudies. "Time and Motion" and "Sleep and Alertness", each conducted at a subset of IM programs and focusing on more detailed data collection at the intern level.

The main protocol will examine patient safety and costs as well as quality of education. The "Time and Motion" substudy examines additional educational outcomes. The "Sleep and Alertness" substudy examines intern sleep time and alertness.

DETAILED DESCRIPTION:
Title: Sleep duration (hours of sleep) as measured with an actigraph Time frame: Measured daily for 14 days

Title: Behavioral alertness as measured with Psychomotor vigilance test Time frame: Measured daily for 14 days

Title: Self perceived sleepiness as measured by the Karolinska Sleepiness Score Time frame: Measured daily for 14 days

Title: Time (hours per day) spent in direct patient care Description: Time spent in direct patient care over 2-4 wks as measured by a trained observer shadowing the intern Time frame: measured daily over 2-4 wks

Title: Trainee satisfaction with education Description: Self-reported satisfaction with education as assessed thru survey questions Time frame: measured at baseline and at end of intervention year

Title: Program director satisfaction with trainee education Description: Self-reported satisfaction with trainee education as assessed thru survey questions Time frame: measured at baseline and end of intervention year

Patient safety and costs:

Title: Total costs of patient care as measured by total Medicare payments Time frame: Measured over year of trial

ELIGIBILITY:
Inclusion Criteria:

* Current internal medicine program in the United States Continued Accreditation status with the ACGME - Program director agrees to:

  1. Randomization to one of the two study arms.
  2. Develop, and share with the study team, institutional duty hour schedules and regulatory policies/procedures that will ensure adherence to, and enforcement of, the duty hour regulations that apply to their study arm
  3. Allow access and analysis of de-identified resident duty hour adherence data/logs, call schedules, and rotation schedules to the Study Team.
  4. Participate, and encourage trainee participation at your institution, in beginning and end of year iCOMPARE surveys.

Exclusion Criteria:

* The investigators excluded 119 programs that comprise the bottom 50% in resident-to-bed ratio and the bottom 25% in patient volume related to the diagnoses by which the patient population will be selected for evaluation of safety outcomes.
* Within the 260 programs that remain, the investigators excluded the 65 in the lowest quartile of program size to ensure we can feasibly obtain sufficient trainee measurements.
* The 195 remaining programs are eligible for inclusion.
* The investigators have also excluded children and VA hospitals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 12 months
  The difference between 30-day mortality rate in the trial year minus the 30-day mortality rate in the pretrial year

SECONDARY OUTCOMES:
Rate of prolonged length of stay | 12 months
  Prolonged length of stay as measured by Medicare data
Total costs of patient care | 12 months
  Total costs of patient care as measured by total Medicare payments
Sleep duration (hours of sleep) | Measured daily for 14 days
  Sleep duration (hours of sleep) as measured with an actigraph
Behavioral alertness | Measured daily for 14 days
  Behavioral alertness as measured with Psychomotor vigilance test
Self perceived sleepiness | Measured daily for 14 days
  Self perceived sleepiness as measured by the Karolinska Sleepiness Score
Time (hours per day) spent in direct patient care | measured daily over 2-4 wks
  Time spent in direct patient care over 2-4 wks as measured by a trained observer shadowing the intern
Trainee satisfaction with education | measured at baseline and at end of intervention year
  Self-reported satisfaction with education as assessed thru survey questions
Program director satisfaction with trainee education | measured at baseline and end of intervention year
  Self-reported satisfaction with trainee education as assessed thru survey questions

CONTACTS AND LOCATIONS:
Overall Officials: David Asch, MD, MBA, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaiyachati KH, Shea JA, Asch DA, Liu M, Bellini LM, Dine CJ, Sternberg AL, Gitelman Y, Yeager AM, Asch JM, Desai SV. Assessment of Inpatient Time Allocation Among First-Year Internal Medicine Residents Using Time-Motion Observations. JAMA Intern Med. 2019 Jun 1;179(6):760-767. doi: 10.1001/jamainternmed.2019.0095. PMID 30985861
- [Derived] Basner M, Asch DA, Shea JA, Bellini LM, Carlin M, Ecker AJ, Malone SK, Desai SV, Sternberg AL, Tonascia J, Shade DM, Katz JT, Bates DW, Even-Shoshan O, Silber JH, Small DS, Volpp KG, Mott CG, Coats S, Mollicone DJ, Dinges DF; iCOMPARE Research Group. Sleep and Alertness in a Duty-Hour Flexibility Trial in Internal Medicine. N Engl J Med. 2019 Mar 7;380(10):915-923. doi: 10.1056/NEJMoa1810641. PMID 30855741
- [Derived] Silber JH, Bellini LM, Shea JA, Desai SV, Dinges DF, Basner M, Even-Shoshan O, Hill AS, Hochman LL, Katz JT, Ross RN, Shade DM, Small DS, Sternberg AL, Tonascia J, Volpp KG, Asch DA; iCOMPARE Research Group. Patient Safety Outcomes under Flexible and Standard Resident Duty-Hour Rules. N Engl J Med. 2019 Mar 7;380(10):905-914. doi: 10.1056/NEJMoa1810642. PMID 30855740
- [Derived] Shea JA, Silber JH, Desai SV, Dinges DF, Bellini LM, Tonascia J, Sternberg AL, Small DS, Shade DM, Katz JT, Basner M, Chaiyachati KH, Even-Shoshan O, Bates DW, Volpp KG, Asch DA; iCOMPARE Research Group. Development of the individualised Comparative Effectiveness of Models Optimizing Patient Safety and Resident Education (iCOMPARE) trial: a protocol summary of a national cluster-randomised trial of resident duty hour policies in internal medicine. BMJ Open. 2018 Sep 21;8(9):e021711. doi: 10.1136/bmjopen-2018-021711. PMID 30244209
- [Derived] Desai SV, Asch DA, Bellini LM, Chaiyachati KH, Liu M, Sternberg AL, Tonascia J, Yeager AM, Asch JM, Katz JT, Basner M, Bates DW, Bilimoria KY, Dinges DF, Even-Shoshan O, Shade DM, Silber JH, Small DS, Volpp KG, Shea JA; iCOMPARE Research Group. Education Outcomes in a Duty-Hour Flexibility Trial in Internal Medicine. N Engl J Med. 2018 Apr 19;378(16):1494-1508. doi: 10.1056/NEJMoa1800965. Epub 2018 Mar 20. PMID 29557719

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT02274818/Prot_SAP_000.pdf